# **STUDY TITLE:**

THE EFFECT OF AN INTERVENTION BASED ON IMPLICIT THEORIES OF PERSONALITY ON
THE PREVENTION OF ADOLESCENT DATING VIOLENCE

# **PROJECT NUMBER:**

PI\_2016\_1\_0023

(Basque Government –Department of education, linguistic policy and culture;

Scientific Policy Administration)

**OCTOBER, 2016** 



#### I. BACKGROUND

Aggressive behavior during adolescence and specifically dating violence are psychosocial problems of crucial clinical and social relevance (Leen et al., 2013; Wincentak, Connolly, & Card, 2017). As children enter adolescence aggressions towards peers give way to other modalities such as dating violence. From a developmental perspective, the first adolescent dating relationships play a relevant role in shaping the general course of development during adolescence, influencing a variety of socioemotional processes and psychological health at this stage, as well as providing an initial platform for the establishment of adult healthy partner relationships (Collins, Welsh, & Furman, 2009; Furman & Shaffer, 2003). Therefore, preventing the development of aggressive behavior towards the partner in adolescence is invaluable. Unfortunately, although there are adequate interventions for preventing dating violence, results for the majority of the previous universal interventions have been poor in terms of behavioral change (Shorey et al., 2012; Whitaker et al., 2006).

The current study will test the efficacy of an Implicit Theory of Personality (ITP) intervention, which has provided excellent results in US both for externalizing problems such as aggressive behavior. Therefore, this study aims to extend this intervention to Spanish adolescents to explore its effect on the prevention of adolescent dating violence. The project includes multiple sources of information: self-reports, parent-reports, and biological data. Thus, the project will contribute from a biopsychosocial and interdisciplinary perspective to the development of universal preventive interventions for intimate partner violence, an important psychological problem in modern societies.

# I.1. Development of aggressive behavior and dating violence

In the last years the rates of aggressive and antisocial behavior have increased in frequency and severity among children and adolescents (Connor, 2012). Although aggressive behavior decreases from childhood to adolescence, more serious forms of violence and deviant behavior tend to peak during this period (Dodge, Coie, & Lynam, 2006). Therefore, adolescence is a period with increased danger of violence and deviant behavior. Furthermore, new forms of aggression (e.g., through new technologies) have emerged and have generated a great deal of attention. Besides, aggressive behavior is persistent over time and predicts later antisocial behavior (Farrington, 2007), thus it is very important to implement preventive interventions at childhood and adolescence.

In particular, dating violence is an important and prevalent problem in adolescence worldwide (Leen et al., 2013; Wincentak et al., 2017). The recent meta-analytic review of teen dating violence prevalence rates by Wincentak and colleagues (2017) showed an overall rate of 20% and 9% for physical and sexual aggression,



respectively. It has been proposed that this high prevalence of adolescent DV is related to the very nature of the developmental period of adolescence, which is characterized by a general pattern of breaking rules and engaging in different types of behaviors that are potentially hazardous to one's health (Fernández-González, O'Leary, & Muñoz-Rivas, 2014; Jessor, 1987; Zweig, Lindberg, & McGinley, 2001). Research on the trajectory of DV throughout adolescence has found that physical partner aggression peaks around the ages of 16 and 17 years (Foshee et al., 2009; Nocentini, Menesini, & Pastorelli, 2010). This peak age of DV during middle-to-late adolescence was also found in Spanish adolescents (Fernández-González et al., 2014). Teen dating relationships are characterized by a lesser level of commitment and a shorter length than romantic relationships in later stages (Wekerle & Wolfe, 1999). However, although at a lower level than in adult life, partner violence may be a moderately steady behavior during adolescence according to the findings of the few longitudinal studies that have examined partner aggression stability in teens (Choi & Temple, 2016; Fritz & Slep, 2009; O'Leary & Slep, 2003). Moreover, adolescents who are involved in violent dating relationships are at a higher risk for a number of psychological, social, academic and physical problems (Chiodo et al., 2012; Choi, Weston, & Temple, 2017; O'Leary, Slep, Avery-Leaf, & Cascardi, 2008).

# I.2. Preventive approaches to aggressive behavior and dating violence

Several aggressive behavior multicomponent interventions with elements directed towards children and adolescents as well as towards their parents and teachers have been developed and have been found to be effective. Some noteworthy examples are the Coping Power (Lochman & Wells, 2002), the Fast Track (Conduct Problems Prevention Research Group, 2002), the Montreal Preventive Treatment Program (Tremblay, Masse, Pagani, & Vitaro, 1996) and the Incredible Years programs (Webster-Stratton, Reid, & Stoolmiller, 2008).

Since the 90s, they have also been developed some programs specifically in the field of dating violence prevention (see for a revision Shorey et al., 2012; Whitaker et al., 2006). Some of the programs are aimed at at-risk populations, as for instance, adolescents that have been victims of child abuse. A noteworthy program in this area is the *Youth Relationships Project* (YRP; Wolfe et al., 2003). The YRP is a program composed of 18 sessions of 120 minutes that uses a health-promotion approach to prevent violence in dating relationships by focusing on positive alternatives to aggression. The intervention was intended for 14–16-year-olds who were considered at-risk of developing abusive dating relationships because of their history of child maltreatment (Wolfe et al., 2003). Universal preventive interventions aimed at the general population of adolescents have also been developed and assessed. Among these prevention programs, some deserve special attention because of their positive results. For instance, the *Safe Dates Project* (Foshee et al., 1998; Foshee et al., 2005)



has been implemented and assessed in a large sample of adolecents in the United States, showing promising results in the prevention of dating violence. However, most of the programs developed until date have shown efficacy in modifying cognitions and attitudes related to dating violence, although behavioral changes have been reported in very few cases. In addition, although these programs have demonstrated to be useful, they are expensive in terms of duration and involvement of various actors (parents, schools, students).

# **Need of universal brief interventions**

In recent years numerous short-term psychosocial interventions have been developed in educational settings with striking effects on several outcomes such as student performance, social integration, and psychological wellbeing (see for a revision Yeager & Walton, 2011). Rigorous field experiments have shown that the effects of such interventions persist for months or even years later. For example, Blackwell, Trzesniewski, and Dweek (2007) got to substantially improve school skills through an intervention based on implicit theories of intelligence, which consisted of showing that intelligence is modifiable and grows when the individual works with effort in challenging tasks. In another intervention, Walton and Cohen (2007, 2011) found that leading students to attribute worries about social integration to the difficulty of the transition to college rather than to students' personal or racial identity can strengthen ethnic minority students' sense of social belonging in school and increase motivation and performance. Furthermore, students who received the intervention reported being happier and healthier in a 3 years posttreatment follow up.

These psychosocial interventions in school can be brief yet impactful because they rely on a rich tradition of research on persuasion and attitude change to powerfully convey psychological ideas (Yeager & Walton, 2011). The crucial elements that contribute to the success of these interventions are the focus on students' experience in school from the students' perspective and the use of impactful delivery mechanisms (Yeager & Walton, 2011). Some of these mechanisms are the following: a) Active role of students, which facilitates deeper message processing; b) Interventions are stealthy. For example, interventions are not presented to the students with the intent to improve performance or other attributes. Thus, students do not feel they are being manipulated so that resistance to intervention is reduced. This approach contributes also to avoid the stigmatization of students. Moreover, the brevity of the interventions also helps to be stealthy. c) Psychosocial interventions have effects over long periods due to recursive processes affecting effects that accumulate over time. Students usually forget the message and the details of the intervention, but this recursive nature triggers other social, psychological and cognitive mechanisms over time.



# Implicit theory of personality (ITP) interventions for emotional and behavioral problems

Recently, Yeager and colleagues have extended this type of brief interventions to prevent emotional and behavioral problems such as depression and aggressive behavior in adolescents. Their approach is based on implicit theories of personality, which refer to the beliefs that people endorse about the malleability of people's socially-relevant traits. An entity theory of personality involves the belief that personal characteristics are fixed and cannot be changed whereas an incremental theory of personality involves the belief that people can change. Past research has found that when adolescents or adults believe that people's traits are fixed and unchangeable, they are more likely to attribute a negative social event (e.g., peer victimization) to their negative traits. They also will tend to infer that the same negative events and other adversities will repeat in the future. Therefore, an entity theory of personality predicts greater shame and negative emotions in adolescents when they cope with stressors such as peer conflicts (Yeager, Trzesniewski, Tirri, Nokelainen, & Dweck, 2011). By the contrary, if adolescents believe that traits can be changed, then their own traits can be improved so that it is unlikely that they become recipients of the same negative events in the future. Furthermore, other people' traits, including those of bullies, can also change. Therefore, the beliefs involved in an incremental theory of personality can be helpful not only for victims but also for perpetrators of bullying. As additional support to this, Rudolph (2010) found that holding an entity theory of peer relationships was associated with a greater tendency to evaluate oneself negatively in the face of peer disapproval and display depressive and aggressive symptoms when victimized.

Yeager and colleagues have developed brief interventions aimed to change entity theories by means of efficient and persuasive intervention tactics that are based on the above mentioned mechanisms. For instance, in one of these interventions, a six-session high school classroom intervention teaching an incremental theory reduced aggressive behavior by 40%, improved depressive symptoms two weeks post-intervention, and increased school attendance (Yeager, Trzesniewski, & Dweck, 2013). Later, they tested the effects of a shorter intervention consisting of only one session. This single session touch an incremental theory via computers. In this session 9<sup>th</sup> grade students read a scientific article about the possibility of personality change, then they read quotes from older students transmitting the same message. Finally, the students wrote a brief essay where they defended the same idea with the aim of transmitting the message to other students in the future. Despite the brevity of this intervention, the results obtained by means of a double-blind randomized experiment showed that it reduced levels of self-reported clinically relevant depression (Miu & Yeager, 2014) and stress levels (Yeager et al., 2014).



#### **II. AIMS AND HYPOTHESES**

The principal aim is to evaluate the effect of an intervention based on Implicit Theories of Personality (ITP) on dating violence in a sample of Spanish adolescents. Grounded on the previous findings obtained in US samples, we will test the efficacy of the ITP intervention by comparing changes in dating violence and from pretreatment to posttreatment and at a six-month and one-year follow up between the group receiving the ITP intervention and a control group that will receive a control educational condition.

Hypothesis: Those adolescents receiving the ITP intervention will show lower frequency of aggressive behavior than the control group after the intervention and at six-month and one-year follow-up.

**A second aim** of this project is to examine whether gender moderates the effects of the intervention in changes in dating violence.

The hypothesis is that the intervention will reduce dating violence involvement in girls than in boys.

#### III. METHODS

This study will use a randomized controlled trial study design with pretest, posttest, six-month follow-up, and one-year follow-up. Group 1 (experimental condition) will receive the ITP intervention and Group 2 (control condition) will receive an educational intervention.

## Study design and participants

We will conduct a double-blind randomized controlled trial (RCT) with two parallel groups in a sample of volunteer adolescents (approximately n=400), and their parents, from several high school centers (ages from 13 to 18 years). The schools will be randomly selected from the Basque Country. Participants will be randomly assigned to the experimental vs control conditions. Group assignation will be done at the individual level within each classroom. Participants were randomized in a 1:1 ratio blocked by gender to one of two groups (experimental versus control condition). They were assigned to their allocated group in class by the researchers.

#### Measures

**Dating violence** will be assessed by means of a self-report questionnaire developed by the research team. Participants who reported having had a dating relationship in the last 6 months (or in the last week at the posttest) will complete a questionnaire to examine dating violence perpetration and victimization. In the first part participants rate the frequency of 25 listed dating aggressive behaviors (perpetration and victimization) in a scale from 0 (never) to 3 (often). Fourteen of the items refer to traditional (face-to-face) dating aggressive acts and 11 items assess acts



of online dating abuse. Specifically, traditional psychological, physical and sexual dating violence included: (1) insulting, (2) threatening to hurt, (3) throwing something at the partner, (4) criticizing the partner in public or private, (5) controlling or trying to prevent with my comments from doing something that I did not want she or he did, (6) attempting to isolate the partner from her or his friends, (7) blaming the partner for problems that were happening or when I got angry, (8) hitting or pulling my partner's hair, (9) discouraging the partner so that he or she does not have hobbies that I do not share, (10) despising or criticizing something that the partner liked, (11) making the partner feel bad for doing something I did not want her or him to do, (12) somehow making it difficult for the partner to go somewhere or talk to someone, (13) kissing or touching the partner against her or his will, and (14) shoving the partner. Items assessing online dating abuse were taken from the Cyber Dating Abuse Questionnaire (Borrajo, Gámez-Guadix, Pereda, & Calvete, 2015) and included: (1) threatening the partner through new technologies to physically harm, (2) creating a fake profile of my partner on a social network to cause problems, (3) using my partner's passwords (phone, social networking, email) to browse, (4) messages and/or contacts without permission, (5) spreading secrets and/or compromised information using new technologies, (6) threatening to spread secrets or embarrassing information using new technologies, (7) using new technologies to pretend to be my partner and create problems for her or him, (8) sending insulting and/or demeaning messages using new technologies, (9) sending and/or posting photos, images and/or videos of my partner with sexual content to other people without permission, (10) using new technologies to control where my partner has been and with whom, (11) spreading rumors, gossip and/or jokes through new technologies with the intention of ridiculing the partner calling excessively to control where the partner was and with whom. Then, only those participants who answer positively any of the previous questions complete a second part of the questionnaire in which they rate the motives and context of the aggression (7 items) and its consequences (5 items). The response choices for each item were defined with the same 4-point scale from 0 (never) to 3 (often).

Parent reports: Parents will be invited to participate by responding measures about their children temperament by means of the revised version of the Early Adolescent Temperament Questionnaire (EATQ-R; Ellis & Rothbart, 2001) and the Big Five Questionnaire for children (BFQ-C; Barbaranelli, Caprara, Rabasca, & Pastorelli, 2003) for parents and depressive symptoms through the CBCL 6/18 (Achenbach, 1991; Achenbach & Edelbrock, 1983). These data will be used in analyses in case that the response rate is enough.

### **Preventive Intervention**

The **ITP intervention** lasts one session (of approximately one hour) and has three main parts: (1) scientific information; (2) normative stories from upperclassmen; and



(3) self-persuasive writing exercise. In the first part, students read a scientific article that provides evidence that individuals have the potential to change. Participants read about actual neurological and behavioral studies showing that behaviors are controlled by "thoughts and feelings in brains," and that pathways in the brain have the potential to be changed under the right circumstances. In the second part, participants read several normative quotes purportedly written by upperclassmen that previously read the same article and endorsed its conclusions. These quotes are obtained from previous interventions and edited by the team. These testimonials are provided to bring credibility to the incremental theory. Finally, in the last part, participants will be asked to write their own version of such a narrative to share with future students, This activity has been shown to facilitate the internalization of the intervention message, building on a long line of research on cognitive dissonance (Walton & Cohen, 2011). For a more complete description of the ITP intervention see Yeager et al. (2013). The intervention will be adapted to the developmental characteristics of the participants.

The **educational intervention** involves scientific information about the human brain. It was designed to be parallel to the experimental intervention and, hence, it has also three main parts. First, participants are asked to read scientific information about the different areas of the brain and their specialties. Second, participants read several testimonials written by upperclassmen about their transition to high school and how their brains help them to adapt to the new space and all the physical differences of the building and the classes. Finally, participants are asked to write a letter to another student explaining the main things he or she has learned about the brain and thinks are important for adapting to the new physical environment in high school. Hence it will control for the possibility that simple optimism about the potential for growth might account for our results. This is a conservative control group. An entity theory control group would be unethical in a longitudinal field experiment because it could teach the belief that personality cannot be changed, which has been associated to negative consequences.

#### **Procedure**

Parental informed consent forms will be sent to parents and adolescents. Those who accept to participate in the study will complete report measures at four waves: (1) one-week before intervention; (2) one-week after intervention; (3) six-months follow-up; and (3) one-year follow-up. Saliva samples will be collected at the same time points. Parents' participants will complete report measures at three waves: (1) one-week before intervention; (2) six-months follow-up; and (3) one-year follow-up. Intervention will be applied one week after the first survey. All the measures will be anonymous and participants will be asked to provide certain data (her/his birth date, first initial of mother's name, and first initial of father's name) to match their questionnaires and intervention tasks over time. Both interventions and assessment



measures will be administered by research assistants during normal class time and last around 50 minutes.

#### **Ethical considerations**

This study aims to develop and implement interventions that will be beneficial for the participating adolescents and other people in the future, by helping to increase their psychological wellbeing. Through randomization, the principle of justice will be respected, allowing all participants to have similar opportunities to receive the intervention. Gender will be considered and similar number of male and female participants will be included in the studies.

The risks are minimal and limited to answering psychological tests on stressors, psychological symptoms and cognitive styles. Previous experience with the same questionnaires indicates that the risk is minimal. Adolescents can also decide to end their participation at any moment. Researchers collecting data will be trained to attend to any difficulty that could emerge while participants are responding to questionnaires. The researchers will give an alternative task (e.g., educational readings) to those participants who decide to end their participation.

Informed consent forms will be sent to parents or legal guardians to complete. Adolescents will also receive written information. The active consent of parents or legal guardians and of adolescents will be necessary for participation in the project. We will incentive adolescents for bringing parent forms, even when decision is negative.

After completing measures, adolescents will be provided with information on services for adolescents (e.g., phone number of attention to adolescents). From an ethical perspective, the most important care aspect is the protection of information. We will follow the Directive 95/46/EC of the European Parliament, *Ley Orgánica 15/99 de 13 de diciembre de Protección de datos de Carácter Personal*, and of the Council of 24 October 1995 on the protection of individuals with regard to the processing of personal data and the free movement of such data. No identification data, such as names or surnames, will be used; instead, we will use a numeric code to match measures across times and sources (parents, and adolescents). Thus, each adolescent, and only he/she, will know his/her code. We will also follow the procedure for data protection that the University of Deusto has registered in the National Data Protection Agency. The project has been approved by the Ethics in Research committee of University of Deusto.

#### IV. STATISTICAL ANALYSES PLAN

Descriptive statistics of sociodemographic and study variables will be provided and several statistical strategies will be used to test the hypotheses. These will include



mixed analyses of variance (ANOVA) and regression analyses. We will employ moderation analyses to test whether sex moderates the effects of the ITV intervention.

#### References

- Achenbach, T. M. (1991). Child Behavior Checklist/4-18 and 1991 profile. *Burlington, Vermont, USA: University of Vermont, Department of Psychiatry*.
- Achenbach, T. M., & Edelbrock, C. S. (1983). Manual for the Child Behavior Checklist/4-18 and revised child behavior profile. *Burlington, Vermont, USA: University of Vermont, Department of Psychiatry*.
- Barbaranelli, C., Caprara, G. V., Rabasca, A., & Pastorelli, C. (2003). A questionnaire for measuring the Big Five in late childhood. *Personality and Individual Differences,* 34(4), 645-664. doi:10.1016/s0191-8869(02)00051-x
- Blackwell, L. S., Trzesniewski, K. H., & Dweck, C. S. (2007). Implicit theories of intelligence predict achievement across an adolescent transition: A longitudinal study and an intervention. Child Development, 78(1), 246-263. doi:10.1111/j.1467-8624.2007.00995.x
- Borrajo, E., Gámez-Guadix, M., Pereda, N., & Calvete, E. (2015). The development and validation of the cyber dating abuse questionnaire among young couples.

  Computers in Human Behavior, 48, 358-365. doi:http://dx.doi.org/10.1016/j.chb.2015.01.063
- Chiodo, D., Crooks, C. V., Wolfe, D. A., McIsaac, C., Hughes, R., & Jaffe, P. G. (2012). Longitudinal prediction and concurrent functioning of adolescent girls demonstrating various profiles of dating violence and victimization. *Prevention Science*, *13*, 350-359. doi: 10.1007/s11121-011-0236-3
- Choi, H. J., & Temple, J. R. (2016). Do gender and exposure to interparental violence moderate the stability of teen dating violence?: Latent transition analysis. *Prevention Science*, 17(3), 367-376. doi: http://dx.doi.org/10.1007/s11121-015-0621-4
- Choi, H. J., Weston, R., & Temple, J. R. (2017). A three-step latent class analysis to identify how different patterns of teen dating violence and psychosocial factors influence mental health. *Journal of Youth and Adolescence, 46,* 854-866. doi: 10.1007/s10964-016-0570-7
- Collins, W. A., Welsh, D. P., & Furman, W. (2009). Adolescent romantic relationships. *Annual Review of Psychology, 60,* 631-652. doi: 10.1146/annurev.psych.60.110707.163459
- Conduct Problems Prevention Research Group. (2002). Using the Fast Track randomized prevention trial to test the early-starter model of the development of serious conduct problems. Development and Psychopathology, 14(4), 925-943. doi:10.1017/s0954579402004133



- Connor, D. F. (2012). Aggression and antisocial behavior in children and adolescents: Research and treatment. New York, USA: Guilford Press.
- Dodge, K. A., Coie, J. D., & Lynam, D. (2006). Aggression and antisocial behavior in youth. In N. Eisenberg (Ed.), Handbook of Child Psychology (6th edition, pp. 719-788). New York, USA: Wiley.
- Ellis, L. K., & Rothbart, M. K. (2001). Revision of the Early Adolescent Temperament Questionnaire. *Biennial Meeting of the Society for Research in Child Development* (2001). Minneapolis, Minnesota, USA.
- Farrington, D. P. (2007). Origins of violent behavior over the life span. In D. J. Flannery, A. T. Vazonyi & I. D. Waldman. (Eds.), The Cambridge handbook of violent behavior and aggression (pp. 19-48). New York, USA: Cambridge University Press.
- Fernández-González, L., O'Leary, K. D., & Muñoz-Rivas, M. J. (2014). Age-related changes in dating aggression in Spanish high school students. *Journal of Interpersonal Violence*, 29, 1132-1152. doi: 10.1177/0886260513506057
- Foshee, V. A., Bauman, K. E., Arriaga, X. B., Helms, R. W., Koch, G. G., y Linder, G. F. (1998). An evaluation of Safe Dates, an adolescent dating violence prevention program. *American Journal of Public Health*, 88, 45-50.
- Foshee, V. A., Bauman, K. E., Ennett, S. T., Suchindran, C., Benefield, T., y Linder, G. F. (2005). Assessing the effects of the dating violence prevention program "Safe Dates" using random coefficient regression modeling. *Prevention Science*, 6, 245-258.
- Foshee, V. A., Benefield, T., Suchindran, C., Ennett, S. T., Bauman, K. E., Karriker-Jaffe, K. J., . . . Mathias, J. (2009). The development of four types of adolescent dating abuse and selected demographic correlates. *Journal of Research on Adolescence*, 19, 380-400. doi: 10.1111/j.1532-7795.2009.00593.x
- Fritz, P. A. T., & Slep, A. M. S. (2009). Stability of physical and psychological adolescent dating aggression across time and partners. *Journal of Clinical Child and Adolescent Psychology*, 38(3), 303-314. doi: 10.1080/15374410902851671
- Furman, W., & Shaffer, L. (2003). The role of romantic relationships in adolescent development. In P. Flosheim (ed.), *Adolescent romantic relations and sexual behavior: Theory, research, and practical implications*, (pp.3-22) Mahwah, NJ, US: Lawrence Erlbaum Associates Publishers.
- Jessor, R. (1987). Problem-behavior theory, psychosocial development, and adolescent problem drinking. *British Journal of Addiction*, 82, 331-342.
- Leen, E., Sorbring, E., Mawer, M., Holdsworth, E., Helsing, B., & Bowen, E. (2013). Prevalence, dynamic risk factors and the efficacy of primary interventions for adolescent dating violence: An international review. *Aggression and Violent Behavior*, 18, 159-174. doi: 10.1016/j.avb.2012.11.015
- Lochman, J. E., & Wells, K. C. (2002). The Coping Power program at the middle-school transition: Universal and indicated prevention effects. Psychology of Addictive Behaviors, 16(4S), S40-S54. doi:10.1037/0893-164x.16.4s.s40



- Miu, A., & Yeager, D. S. (2014). Preventing symptoms of depression by teaching adolescents that people can change: Effects of a brief incremental theory of personality intervention at 9-month follow-up. Clinical Psychological Science, 3(5), 726-743. doi:10.1177/2167702614548317
- Nocentini, A., Menesini, E., & Pastorelli, C. (2010). Physical dating aggression growth during adolescence. *Journal of Abnormal Child Psychology, 38*, 353-365. doi: 10.1007/s10802-009-9371-8
- O'Leary, K. D., & Slep, A. M. S. (2003). A dyadic longitudinal model of adolescent dating aggression. *Journal of Clinical Child and Adolescent Psychology*, 32(3), 314-327.
- O'Leary, K. D., Slep, A. M. S., Avery-Leaf, S., & Cascardi, M. (2008). Gender differences in dating aggression among multiethnic high school students. *Journal of Adolescent Health*, 42, 473-479. doi: 10.1016/j.jadohealth.2007.09.012
- Rudolph, K. D. (2010). Implicit theories of peer relationships. Social Development, 19(1), 113-129. doi:10.1111/j.1467-9507.2008.00534.x
- Shorey, R. C., Zucosky, H., Brasfield, H., Febres, J., Cornelius, T. L., Sage, C., y Stuart, G. L. (2012). Dating violence prevention programming: Directions for future interventions. *Aggression and Violent Behavior*, *17*, 289-296.
- Tremblay, R. E., Masse, L., Pagani, L., & Vitaro, F. (1996). From childhood physical aggression to adolescent maladjustment: The Montreal Prevention Experiment. In R. D. Peters & R. J. McMahon. (Eds.), Preventing childhood disorders, substance abuse, and delinquency (pp. 268-298). Thousand Oaks, California, USA: Sage Publications.
- Walton, G. M., & Cohen, G. L. (2007). A question of belonging: Race, social fit, and achievement. Journal of Personality and Social Psychology, 92(1), 82-96. doi:10.1037/0022-3514.92.1.82
- Walton, G. M., & Cohen, G. L. (2011). A brief social-belonging intervention improves academic and health outcomes of minority students. Science, 331(6023), 1447-1451. doi:10.1126/science.1198364
- Webster-Stratton, C., Reid, J., & Stoolmiller, M. (2008). Preventing conduct problems and improving school readiness: Evaluation of the Incredible Years Teacher and Child Training Programs in high-risk schools. Journal of Child Psychology and Psychiatry, 49(5), 471-88. doi:10.1111/j.1469-7610.2007.01861.x
- Wekerle, C., & Wolfe, D. A. (1999). Dating violence in mid-adolescence: Theory, significance, and emerging prevention initiatives. *Clinical Psychology Review*, 19, 435-456.
- Whitaker, D. J., Morrison, S., Lindquist, C., Hawkins, S. R., O'Neil, J. A., Nesius, A. M., ... Reese, L. R. (2006). A critical review of interventions for the primary prevention of perpetration of partner violence. *Aggression and Violent Behavior, 11*, 151-166.



- Wincentak, K., Connolly, J., & Card, N. (2017). Teen dating violence: A meta-analytic review of prevalence rates. *Psychology of Violence*, *7*, 224-241. doi: 10.1037/a0040194
- Wolfe, D. A., Wekerle, C., Scott, K., Straatman, A.-L., Grasley, C., y Reitzel-Jaffe, D. (2003). Dating violence prevention with at-risk youth: A controlled outcome evaluation. *Journal of Consulting and Clinical Psychology*, 71, 279-291.
- Yeager, D. S., & Walton, G. M. (2011). Social-psychological interventions in education: They're not magic. Review of Educational Research, 81(2), 267-301. doi:10.3102/0034654311405999
- Yeager, D. S., Trzesniewski, K., & Dweck, C. S. (2013). An implicit theories of personality intervention reduces adolescent aggression in response to victimization and exclusion. Child Development, 84(3), 970-988. doi:10.1111/cdev.12003
- Yeager, D. S., Trzesniewski, K., Tirri, K., Nokelainen, P., & Dweck, C. S. (2011). Adolescents' implicit theories predict desire for vengeance: Correlational and experimental evidence. Developmental Psychology, 47(4), 1090-1107. doi:10.1037/a0023769
- Yeager, D.S., Johnson, R., Spitzer, B., Trzesniewski, K., Powers, J., & Dweck, C.S. (2014). The far-reaching effects of believing people can change: Implicit theories of personality shape stress, health, and achievement during adolescence. Journal of Personality and Social Psychology, 106(6), 867-884. doi:10.1037/a0036335
- Zweig, J. M., Lindberg, L. D., & McGinley, K. A. (2001). Adolescent health risk profiles: The co-occurrence of health risks among females and males. *Journal of Youth and Adolescence*, *30*, 707-728. doi: 10.1023/a:1012281628792